CLINICAL TRIAL: NCT06099028
Title: Heart Failure Treatment Pattern Analysis of HF Patients in HF Centers and Non-HF Centers in China: a Retrospective Database-based Study
Brief Title: Heart Failure Treatment Pattern Analysis of HF Patients in HF Centers and Non-HF Centers in China
Status: Completed | Type: Observational
Sponsor: Peking University First Hospital (Other)
Collaborators: China Cardiovascular Association (Other); AstraZeneca (Industry)
Responsible Party: Principal Investigator, Yong Huo, Prof, Peking University First Hospital
Other Study IDs: ESR-22-22035
Record Dates: First submitted 2023-09-17; First posted 2023-10-25 (Actual); Last update posted 2024-01-23 (Actual); Status verified 2024-01

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- HF center: heart failure patients enrolled from heart failure center hospitals
  Interventions: Other: no intervention
- non-HF center: heart failure patients enrolled from non-heart failure center hospitals

INTERVENTIONS:
Other: no intervention — no intervention
  Groups: HF center

SUMMARY:
This is a retrospective, researcher-initiated, database-based study that will retrospectively observe the treatment and medication patterns of about 22,500 patients with heart failure from 25 heart failure centers and 25 non-heart failure centers in the database of heart failure center. The proportion of patients with heart failure treatment drugs reaching the target dose recommended in the guidelines and discontinuation rate will be observed at 1 month, 3 months and 12 months follow up time point. The purpose of this study is to illustrate the current HF treatment status in HF center hospitals and non-HF center hospitals, which may provide insights for improving the clinical practice of heart failure treatment in China, and promote the standardization of heart failure treatment in China.

ELIGIBILITY:
Inclusion Criteria:

* An index HF diagnosis date in the records
* Age ≥ 18 years old at initial diagnosis date
* HF patients baseline characteristic record

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will include HF patients extracted from the HF centers Database. The enrolment of HF cases was via the consecutive sampling. In this study, the study time frame is from 2021.09 to 2023.03. The index date will be defined as the discharge date after the first HF admission (inpatient) record shown in the database, (i.e., the discharge date is the date entry into the HF centers Database). Given that previous treatment condition of these patients before the enrolment in this database is unknown, the baseline information was only collected at the index date. Patient follow-ups were scheduled at 1 month, 3 months and 12 months after the first discharge. The window of follow-up was set for ±14 days.
Sampling Method: Non-Probability Sample
Enrollment: 22500 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2023-03-31 (Actual); Study Completion 2023-03-31 (Actual)

PRIMARY OUTCOMES:
Number of GDMT drugs (classified as RAASi (including ARNI), beta blockers, MRA and SGLT2i) | At baseline and at 1 month, 3 month, 12 month follow-up time point
  Numbers of GDMT drugs of HF patients stratified by HF ejection fraction and by HF Center and Non-HF Center
Use rates of GDMT drugs | At baseline and at 1 month, 3 month, 12 month follow-up time point
  The percentage of patients using each GDMT drug，stratified by HF ejection fraction and by HF Center and Non-HF Center

SECONDARY OUTCOMES:
The proportion of patients using 2 types of GDMT drugs | At baseline and at 1 month, 3 month, 12 month follow-up time point
  The percentage of patients using 2 of any 4 GDMT drugs，stratified by HF ejection fraction and by HF Center and Non-HF Center
The proportion of patients using 3 types of GDMT drugs | At baseline and at 1 month, 3 month, 12 month follow-up time point
  The percentage of patients using 3 of any 4 GDMT drugs，stratified by HF ejection fraction and by HF Center and Non-HF Center
The proportion of patients using 4 types of GDMT drugs | At baseline and at 1 month, 3 month, 12 month follow-up time point
  The percentage of patients using all types of GDMT drugs，stratified by HF ejection fraction and by HF Center and Non-HF Center
The proportion of patients with each GDMT drug in the target dose | at 1 month, 3 month, 12 month follow-up time point
  The percentage of patients who achieved the target dose of each GDMT drug, stratified by HF ejection fraction and by HF Center and Non-HF Center
Discontinuation rate of each GDMT drug | at 1 month, 3 month, 12 month follow-up time point
  The percentage of patients who discontinued GDMT drugs, stratified by HF ejection fraction and by HF Center and Non-HF Center

CONTACTS AND LOCATIONS:
Overall Officials: Huo Yong, MD., Principal Investigator — Peking University First Hospital
Locations (1):
- Department of Cardiology, Peking University First Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] GBD 2017 Disease and Injury Incidence and Prevalence Collaborators. Global, regional, and national incidence, prevalence, and years lived with disability for 354 diseases and injuries for 195 countries and territories, 1990-2017: a systematic analysis for the Global Burden of Disease Study 2017. Lancet. 2018 Nov 10;392(10159):1789-1858. doi: 10.1016/S0140-6736(18)32279-7. Epub 2018 Nov 8. PMID 30496104
- [Background] Cowie MR, Anker SD, Cleland JGF, Felker GM, Filippatos G, Jaarsma T, Jourdain P, Knight E, Massie B, Ponikowski P, Lopez-Sendon J. Improving care for patients with acute heart failure: before, during and after hospitalization. ESC Heart Fail. 2014 Dec;1(2):110-145. doi: 10.1002/ehf2.12021. Epub 2015 Jan 21. PMID 28834628
- [Background] Groenewegen A, Rutten FH, Mosterd A, Hoes AW. Epidemiology of heart failure. Eur J Heart Fail. 2020 Aug;22(8):1342-1356. doi: 10.1002/ejhf.1858. Epub 2020 Jun 1. PMID 32483830
- [Background] Jones NR, Roalfe AK, Adoki I, Hobbs FDR, Taylor CJ. Survival of patients with chronic heart failure in the community: a systematic review and meta-analysis. Eur J Heart Fail. 2019 Nov;21(11):1306-1325. doi: 10.1002/ejhf.1594. Epub 2019 Sep 16. PMID 31523902
- [Background] Setoguchi S, Stevenson LW, Schneeweiss S. Repeated hospitalizations predict mortality in the community population with heart failure. Am Heart J. 2007 Aug;154(2):260-6. doi: 10.1016/j.ahj.2007.01.041. PMID 17643574
- [Background] Bottle A, Kim D, Aylin P, Cowie MR, Majeed A, Hayhoe B. Routes to diagnosis of heart failure: observational study using linked data in England. Heart. 2018 Apr;104(7):600-605. doi: 10.1136/heartjnl-2017-312183. Epub 2017 Oct 5. PMID 28982720
- [Background] Lawson CA, Zaccardi F, Squire I, Ling S, Davies MJ, Lam CSP, Mamas MA, Khunti K, Kadam UT. 20-year trends in cause-specific heart failure outcomes by sex, socioeconomic status, and place of diagnosis: a population-based study. Lancet Public Health. 2019 Aug;4(8):e406-e420. doi: 10.1016/S2468-2667(19)30108-2. PMID 31376859
- [Background] Ghazi L, Yamamoto Y, Riello RJ, Coronel-Moreno C, Martin M, O'Connor KD, Simonov M, Huang J, Olufade T, McDermott J, Dhar R, Inzucchi SE, Velazquez EJ, Wilson FP, Desai NR, Ahmad T. Electronic Alerts to Improve Heart Failure Therapy in Outpatient Practice: A Cluster Randomized Trial. J Am Coll Cardiol. 2022 Jun 7;79(22):2203-2213. doi: 10.1016/j.jacc.2022.03.338. Epub 2022 Apr 3. PMID 35385798
- [Background] McDonagh TA, Metra M, Adamo M, Gardner RS, Baumbach A, Bohm M, Burri H, Butler J, Celutkiene J, Chioncel O, Cleland JGF, Coats AJS, Crespo-Leiro MG, Farmakis D, Gilard M, Heymans S, Hoes AW, Jaarsma T, Jankowska EA, Lainscak M, Lam CSP, Lyon AR, McMurray JJV, Mebazaa A, Mindham R, Muneretto C, Francesco Piepoli M, Price S, Rosano GMC, Ruschitzka F, Kathrine Skibelund A; ESC Scientific Document Group. 2021 ESC Guidelines for the diagnosis and treatment of acute and chronic heart failure. Eur Heart J. 2021 Sep 21;42(36):3599-3726. doi: 10.1093/eurheartj/ehab368. No abstract available. PMID 34447992
- [Background] Heidenreich PA, Bozkurt B, Aguilar D, Allen LA, Byun JJ, Colvin MM, Deswal A, Drazner MH, Dunlay SM, Evers LR, Fang JC, Fedson SE, Fonarow GC, Hayek SS, Hernandez AF, Khazanie P, Kittleson MM, Lee CS, Link MS, Milano CA, Nnacheta LC, Sandhu AT, Stevenson LW, Vardeny O, Vest AR, Yancy CW. 2022 AHA/ACC/HFSA Guideline for the Management of Heart Failure: A Report of the American College of Cardiology/American Heart Association Joint Committee on Clinical Practice Guidelines. J Am Coll Cardiol. 2022 May 3;79(17):e263-e421. doi: 10.1016/j.jacc.2021.12.012. Epub 2022 Apr 1. PMID 35379503